CLINICAL TRIAL: NCT04970485
Title: Evaluation of the Talking Matters Teen Pregnancy Prevention Program Through a Randomized Controlled Trial Design
Brief Title: Evaluation of the Talking Matters Teen Pregnancy Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Public Health Management Corporation (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Archana LaPollo, Senior Project Director, Public Health Management Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2003
Record Dates: First submitted 2021-01-11; First posted 2021-07-21 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Pregnancy in Adolescence

STUDY DESIGN:
Intervention Model Description: Individual randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Talking Matters intervention (Experimental): Talking Matters is a group-level, two-pronged intervention for Black and African American 14 to 19 year old adolescents recruited from school- and community-based settings in Philadelphia, PA. Goals are to reduce teens' risk for unplanned pregnancy, sexually transmitted infections, and HIV, and to strengthen protective factors to improve health. The two prongs include (1) an adolescent-focused five-session, group-level intervention called We Get to Choose (WGTC) covering sexual and reproductive health (SRH) knowledge and skills, decision making and self-worth, healthy relationships, substance use and mental health; and (2) an adult-focused three-session, group-level training called Let's Talk Real Talk (LTRT) to build SRH knowledge and skills to communicate with teens about SRH. An opportunity to connect WGTC participants to trusted adults who completed LTRT is provided during one facilitated session conducted each quarter. LTRT participants are not human subjects of the study.
  Interventions: Behavioral: Talking Matters
- Control Group (No Intervention): Business as usual

INTERVENTIONS:
Behavioral: Talking Matters — Group-level, facilitator-led behavioral intervention for 14-19 year old Black and African American adolescents with an intergenerational component to reduce teen pregnancy, strengthen protective factors to improve optimal health, and increase access to trusted adults.
  Other Names: We Get to Choose; Let's Talk Real Talk
  Arms: Talking Matters intervention

SUMMARY:
A culturally tailored program that creates a safe, open space to increase knowledge, self-efficacy, skills, and comfort related to sexual and reproductive health, including HIV/STI and teen pregnancy prevention, mental health, and substance use risk reduction behavior, and strengthens protective factors, decision-making skills, and connections to trusted adults may help participants chart a path toward optimal health. To address a significant gap in evidence-based, culturally-tailored sexual and reproductive health services for Black and African American adolescents, Public Health Management Corporation (PHMC) is conducting a rigorous evaluation of an innovative group-level, two pronged intervention called Talking Matters using an individual randomized control trial (RCT) design. Due to social distancing guidelines during COVID-19 at the start of the study, all Talking Matters activities, including recruitment, screening, consent, intervention implementation, and data collection, will be conduct virtually and remotely.

Developed and piloted over the past two years through FY2018 Phase I New and Innovative Strategies (Tier 2) to Prevent Teen Pregnancy and Promote Healthy Adolescence funding from the Office of Population Affairs (OPA), Talking Matters is a promising group-level, two-pronged intervention tailored for urban Black and African American 14 to 19 year old adolescents who are recruited from school- and community-based settings in Philadelphia, PA. Grounded in Social Cognitive Theory, the Transtheoretical Model, and Self-Determination Theory, and using evidence-based Motivational Interviewing strategies, the primary goals of Talking Matters are to reduce adolescents' risk for teen and unplanned pregnancy, sexually transmitted infections (STIs) and HIV, and to strengthen protective factors improve optimal health.

The two prongs of Talking Matters include (1) an adolescent-focused five-session, group-level intervention called We Get to Choose (WGTC) and (2) an adult-focused three-session, group-level training called Let's Talk Real Talk (LTRT). An opportunity to connect WGTC participants to trusted adults who completed LTRT is provided during one facilitated session conducted each quarter. Adult participants of the LTRT training are not human subjects of the Talking Matters study.

ELIGIBILITY:
Inclusion Criteria:

* Identifies as Black or African American
* 14 to 19 years old at baseline
* Lives in Philadelphia, PA
* English-speaking
* Able to or will be able to obtain access to the internet through a phone, tablet, or computer

Exclusion Criteria:

* Does not identify as Black or African American
* Less than 14 years old or 20 years or older at baseline
* Does not live in Philadelphia, PA
* Unable to speak or understand English
* Unable to access internet through a phone, tablet, or computer

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 321 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in the number of oral, vaginal, and/or anal sex episodes without a condom, female condom, or dental dam in the past 60 days (2 months) from baseline to follow up. | Baseline up to 3 months post-baseline
Change in the number of oral, vaginal, and/or anal sex episodes without a condom, female condom, or dental dam in the past 60 days (2 months) from baseline to follow up. | Baseline up to 6 months post-baseline
Change in the number of vaginal sex episodes without any form of contraception (including condoms) in the past 60 days (2 months) from baseline to follow up. | Baseline up to 3 months post-baseline
Change in the number of vaginal sex episodes without any form of contraception (including condoms) in the past 60 days (2 months) from baseline to follow up. | Baseline up to 6 months post-baseline
Change in the number of partners with whom participants had oral, vaginal, and/or anal sex without a condom, female condom, or dental dam in the past 60 days (2 months) from baseline to follow up. | Baseline up to 3 months post-baseline
Change in the number of partners with whom participants had oral, vaginal, and/or anal sex without a condom, female condom, or dental dam in the past 60 days (2 months) from baseline to follow up. | Baseline up to 6 months post-baseline
Maintained condom use at last vaginal sex (yes/no) from baseline to follow up. | Baseline up to 3 months post-baseline
Change in condom use at last vaginal sex (yes/no) from baseline to follow up. | Baseline up to 3 months post-baseline
Maintained condom use at last vaginal sex (yes/no) from baseline to follow up. | Baseline up to 6 months post-baseline
Change in condom use at last vaginal sex (yes/no) from baseline to follow up. | Baseline up to 6 months post-baseline
Change in self-efficacy for communicating with sexual partners about sexual and reproductive health from baseline to follow up. | Baseline up to 5 weeks post-baseline
  Abbreviated Sexual communication self-efficacy scales from The sexual communication self-efficacy scale and Canadian Sexual Health Indicators Survey-Pilot Test And Validation Phase: Final Technical Report.
  Centre for Communicable Diseases and Infection Control, Infectious Disease Prevention and Control Branch, Public Health Agency of Canada, 2012. (16 of 20 items used)
Change in self-efficacy for communicating with sexual partners about sexual and reproductive health from baseline to follow up. | Baseline up to 3 months post-baseline
  Abbreviated Sexual communication self-efficacy scales from The sexual communication self-efficacy scale and Canadian Sexual Health Indicators Survey-Pilot Test And Validation Phase: Final Technical Report.
  Centre for Communicable Diseases and Infection Control, Infectious Disease Prevention and Control Branch, Public Health Agency of Canada, 2012. (16 of 20 items used)
Change in self-efficacy for communicating with sexual partners about sexual and reproductive health from baseline to follow up. | Baseline up to 6 months post-baseline
  Abbreviated Sexual communication self-efficacy scales from The sexual communication self-efficacy scale and Canadian Sexual Health Indicators Survey-Pilot Test And Validation Phase: Final Technical Report.
  Centre for Communicable Diseases and Infection Control, Infectious Disease Prevention and Control Branch, Public Health Agency of Canada, 2012. (16 of 20 items used)

SECONDARY OUTCOMES:
Change in sexual and reproductive health knowledge from baseline to follow up. | Baseline up to 5 weeks post-baseline
  As measured by the number of correct items reported on a 22-item questionnaire comprising modified items from Sexual Transmitted Diseases Knowledge Questionnaire (Jaworski, B. C., & Carey, M. P. (2007). Development and psychometric evaluation of a self-administered questionnaire to measure knowledge of sexually transmitted diseases. AIDS and Behavior, 11(4), 557-574); items from Anderman, E. M., Cupp, P. K., Lane, D. R., Zimmerman, R., Gray, D. L., & O'Connell, A. (2011). Classroom goal structures and HIV and pregnancy prevention education in rural high school health classrooms. Journal of Research on Adolescence, 21(4), 904-922; Section 7 from Cleland, J. (2001). Illustrative questionnaire for interview-surveys with young people. Asking Young People About Sexual and Reproductive Behaviors. Illustrative Core Instruments, Geneva: World Health Organization.
Change in sexual and reproductive health knowledge from baseline to follow up. | Baseline up to 3 months post-baseline
  As measured by the number of correct items reported on a 22-item questionnaire comprising modified items from Sexual Transmitted Diseases Knowledge Questionnaire (Jaworski, B. C., & Carey, M. P. (2007). Development and psychometric evaluation of a self-administered questionnaire to measure knowledge of sexually transmitted diseases. AIDS and Behavior, 11(4), 557-574); items from Anderman, E. M., Cupp, P. K., Lane, D. R., Zimmerman, R., Gray, D. L., & O'Connell, A. (2011). Classroom goal structures and HIV and pregnancy prevention education in rural high school health classrooms. Journal of Research on Adolescence, 21(4), 904-922; Section 7 from Cleland, J. (2001). Illustrative questionnaire for interview-surveys with young people. Asking Young People About Sexual and Reproductive Behaviors. Illustrative Core Instruments, Geneva: World Health Organization.
Change in sexual and reproductive health knowledge from baseline to follow up. | Baseline up to 6 months post-baseline
  As measured by the number of correct items reported on a 22-item questionnaire comprising modified items from Sexual Transmitted Diseases Knowledge Questionnaire (Jaworski, B. C., & Carey, M. P. (2007). Development and psychometric evaluation of a self-administered questionnaire to measure knowledge of sexually transmitted diseases. AIDS and Behavior, 11(4), 557-574); items from Anderman, E. M., Cupp, P. K., Lane, D. R., Zimmerman, R., Gray, D. L., & O'Connell, A. (2011). Classroom goal structures and HIV and pregnancy prevention education in rural high school health classrooms. Journal of Research on Adolescence, 21(4), 904-922; Section 7 from Cleland, J. (2001). Illustrative questionnaire for interview-surveys with young people. Asking Young People About Sexual and Reproductive Behaviors. Illustrative Core Instruments, Geneva: World Health Organization.
Change in knowledge, expectations, and attitudes about healthy relationships from baseline to follow up. | Baseline up to 5 weeks post-baseline
  Abbreviated Healthy Relationship Knowledge, Expectations, and Attitudes domain from the Health Marriage and Relationship Education Models and Measures Project.(Scott, M.E., Moore, K.A., Fish, H., Benedetti, A., & Erikson, S. (2015). Healthy marriage and relationship education: Recommended outcome measures for adolescents. OPRE Report #2015-65a. Prepared by Child Trends. Washington, DC: Office of Planning, Research and Evaluation, Administration for Children and Families, U.S. Department of Health and Human Services.)
Change in knowledge, expectations, and attitudes about healthy relationships from baseline to follow up. | Baseline up to 3 months post-baseline
  Abbreviated Healthy Relationship Knowledge, Expectations, and Attitudes domain from the Health Marriage and Relationship Education Models and Measures Project.(Scott, M.E., Moore, K.A., Fish, H., Benedetti, A., & Erikson, S. (2015). Healthy marriage and relationship education: Recommended outcome measures for adolescents. OPRE Report #2015-65a. Prepared by Child Trends. Washington, DC: Office of Planning, Research and Evaluation, Administration for Children and Families, U.S. Department of Health and Human Services.)
Change in knowledge, expectations, and attitudes about healthy relationships from baseline to follow up. | Baseline up to 6 months post-baseline
  Abbreviated Healthy Relationship Knowledge, Expectations, and Attitudes domain from the Health Marriage and Relationship Education Models and Measures Project.(Scott, M.E., Moore, K.A., Fish, H., Benedetti, A., & Erikson, S. (2015). Healthy marriage and relationship education: Recommended outcome measures for adolescents. OPRE Report #2015-65a. Prepared by Child Trends. Washington, DC: Office of Planning, Research and Evaluation, Administration for Children and Families, U.S. Department of Health and Human Services.)
Change in mental health literacy from baseline to follow up. | Baseline up to 5 weeks post-baseline
  18 items scored from 1 to 4 (higher score=higher knowledge) from O'Connor, M., & Casey, L. (2015). The Mental Health Literacy Scale (MHLS): A new scale-based measure of mental health literacy. Psychiatry research, 229(1-2), 511-516. and Self efficacy for stress management from Hansen, W. B., & McNeal Jr, R. B. (1997). How DARE works: An examination of program effects on mediating variables. Health education & behavior, 24(2), 165-176.
Change in mental health literacy from baseline to follow up. | Baseline up to 3 months post-baseline
  18 items scored from 1 to 4 (higher score=higher knowledge) from O'Connor, M., & Casey, L. (2015). The Mental Health Literacy Scale (MHLS): A new scale-based measure of mental health literacy. Psychiatry research, 229(1-2), 511-516. and Self efficacy for stress management from Hansen, W. B., & McNeal Jr, R. B. (1997). How DARE works: An examination of program effects on mediating variables. Health education & behavior, 24(2), 165-176.
Change in mental health literacy from baseline to follow up. | Baseline up to 6 months post-baseline
  18 items scored from 1 to 4 (higher score=higher knowledge) from O'Connor, M., & Casey, L. (2015). The Mental Health Literacy Scale (MHLS): A new scale-based measure of mental health literacy. Psychiatry research, 229(1-2), 511-516. and Self efficacy for stress management from Hansen, W. B., & McNeal Jr, R. B. (1997). How DARE works: An examination of program effects on mediating variables. Health education & behavior, 24(2), 165-176.
Change in intentions to use condoms from baseline to follow up. | Baseline up to 5 weeks post-baseline
  Sakeah, J. K. (2017). Determinants of Condom use intentions among University students in Ghana (Doctoral dissertation, Lethbridge, Alta: University of Lethbridge, Faculty of Health Sciences).
Change in intentions to use condoms from baseline to follow up. | Baseline up to 3 months post-baseline
  Sakeah, J. K. (2017). Determinants of Condom use intentions among University students in Ghana (Doctoral dissertation, Lethbridge, Alta: University of Lethbridge, Faculty of Health Sciences).
Change in intentions to use condoms from baseline to follow up. | Baseline up to 6 months post-baseline
  Sakeah, J. K. (2017). Determinants of Condom use intentions among University students in Ghana (Doctoral dissertation, Lethbridge, Alta: University of Lethbridge, Faculty of Health Sciences).
Change in self-efficacy for communicating with trusted adults about sexual and reproductive health from baseline to follow up | Baseline up to 5 weeks post-baseline
  Modified Parent-Teen Communication About Premarital Sex from Jaccard, J., Dittus, P. J., & Gordon, V. V. (2000). Parent-teen communication about premarital sex: Factors associated with the extent of communication. Journal of Adolescent Research, 15(2), 187-208.
Change in self-efficacy for communicating with trusted adults about sexual and reproductive health from baseline to follow up | Baseline up to 3 months post-baseline
  Modified Parent-Teen Communication About Premarital Sex from Jaccard, J., Dittus, P. J., & Gordon, V. V. (2000). Parent-teen communication about premarital sex: Factors associated with the extent of communication. Journal of Adolescent Research, 15(2), 187-208.
Change in self-efficacy for communicating with trusted adults about sexual and reproductive health from baseline to follow up | Baseline up to 6 months post-baseline
  Modified Parent-Teen Communication About Premarital Sex from Jaccard, J., Dittus, P. J., & Gordon, V. V. (2000). Parent-teen communication about premarital sex: Factors associated with the extent of communication. Journal of Adolescent Research, 15(2), 187-208.
Change in self-efficacy for using condoms from baseline to follow up. | Baseline up to 5 weeks post-baseline
  Abbreviated condom use self-efficacy scale from Asante, K. O., & Doku, P. N. (2010). Cultural adaptation of the condom use self efficacy scale (CUSES) in Ghana. BMC public health, 10(1), 1-7. (12 of 14 items used)
Change in self-efficacy for using condoms from baseline to follow up. | Baseline up to 3 months post-baseline
  Abbreviated condom use self-efficacy scale from Asante, K. O., & Doku, P. N. (2010). Cultural adaptation of the condom use self efficacy scale (CUSES) in Ghana. BMC public health, 10(1), 1-7. (12 of 14 items used)
Change in self-efficacy for using condoms from baseline to follow up. | Baseline up to 6 months post-baseline
  Abbreviated condom use self-efficacy scale from Asante, K. O., & Doku, P. N. (2010). Cultural adaptation of the condom use self efficacy scale (CUSES) in Ghana. BMC public health, 10(1), 1-7. (12 of 14 items used)
Change in attitudes and beliefs about healthy decision making around risk reduction behaviors from baseline to follow up | Baseline up to 5 weeks post-baseline
  Abbreviated Making Decisions in Everyday life instrument. from Mincemoyer, C., Perkins, D. F., & Munyua, C. (2005). Measuring the impact of youth development programs: A national on-line youth life skills evaluation system. In The Forum for Family and Consumer Issues (Vol. 10, No. 2).
Change in attitudes and beliefs about healthy decision making around risk reduction behaviors from baseline to follow up | Baseline up to 3 months post-baseline
  Abbreviated Making Decisions in Everyday life instrument. from Mincemoyer, C., Perkins, D. F., & Munyua, C. (2005). Measuring the impact of youth development programs: A national on-line youth life skills evaluation system. In The Forum for Family and Consumer Issues (Vol. 10, No. 2).
Change in attitudes and beliefs about healthy decision making around risk reduction behaviors from baseline to follow up | Baseline up to 6 months post-baseline
  Abbreviated Making Decisions in Everyday life instrument. from Mincemoyer, C., Perkins, D. F., & Munyua, C. (2005). Measuring the impact of youth development programs: A national on-line youth life skills evaluation system. In The Forum for Family and Consumer Issues (Vol. 10, No. 2).

CONTACTS AND LOCATIONS:
Overall Officials: Archana B LaPollo, MPH, Principal Investigator — Public Health Management Corporation
Locations (1):
- Public Health Management Corporation, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No